CLINICAL TRIAL: NCT06225167
Title: Pharmacist-Driven Stress Ulcer Prophylaxis Minimization in the Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 005.PHA.2023.R
Record Dates: First submitted 2023-07-06; First posted 2024-01-25 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-01

CONDITIONS: Stress Ulcer
MeSH Terms: conditions — Duodenal Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Protocol Group: Patients will be analyzed during the time frame of February 2020 to February 2023 for the protocol group
  Interventions: Behavioral: To evaluate the effectiveness and safety of a pharmacist-driven protocol to discontinue stress ulcer prophylaxis in ICU patients when it is no longer indicated according to pre-defined criteria.
- Non Protocol Group: Patients will be analyzed during the time frame of February 2017 to February 2020 for the non-protocol group.
  Interventions: Behavioral: To evaluate the effectiveness and safety of a pharmacist-driven protocol to discontinue stress ulcer prophylaxis in ICU patients when it is no longer indicated according to pre-defined criteria.

INTERVENTIONS:
Behavioral: To evaluate the effectiveness and safety of a pharmacist-driven protocol to discontinue stress ulcer prophylaxis in ICU patients when it is no longer indicated according to pre-defined criteria. — To evaluate the effectiveness and safety of a pharmacist-driven protocol to discontinue stress ulcer prophylaxis in ICU patients when it is no longer indicated according to pre-defined criteria.
  To compare the incidence of overt GI bleeds (defined as hematemesis, bloody nasogastric tube aspirate, or melena) between patients who were on stress ulcer prophylaxis versus patients whose acid suppression therapy was discontinued through the stress ulcer prophylaxis minimization protocol.

SUMMARY:
Pharmacologic stress ulcer prophylaxis is routinely used in the intensive care unit (ICU) to prevent upper gastrointestinal (GI) bleeding in critically ill patients.

DETAILED DESCRIPTION:
Historically, the two independent risk factors for stress-related GI bleeds were coagulopathy and mechanical ventilation for more than 48 hours; however, several additional risk factors have been identified, such as shock, multiple organ failure, traumatic brain injury, and major burns.

Acid suppressive medications such as proton pump inhibitors or histamine-2 receptor antagonists are prescribed to reduce the rate of bleeding from stress ulceration despite a lack of benefit from placebo-controlled trials. In addition to lack of proven benefit, the incidence of clinically significant stress-related GI bleeding has decreased over time, likely due to improvements in critical care and earlier enteral feeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years ICU location status

Exclusion Criteria:

* If patient has one of the following:

  * Coagulopathy (defined as: platelets < 50,000/µL, international normalized ratio(INR) > 1.5, or partial thromboplastin time > 2 times the control value)
  * Mechanical ventilation for > 48 hours and on < 50% goal tube feeds
  * Shock state on vasopressors/inotropes and on < 50% goal tube feeds (or < 50% of diet)
  * On total parenteral nutrition
  * Use of acid suppressive therapy prior to admission
  * Admission with GI bleeding
  * History of peptic ulcer disease
  * Surgery on the GI tract or cardiac surgery during the current hospital admission
  * Pregnancy
  * H. pylori infection treatment
  * Hypersecretory disorder (ex: Zollinger-Ellison)
  * Known erosive esophagitis/gastritis (not heartburn or gastroesophageal reflux disease)
  * Traumatic brain injury with Glasgow Coma Scale score ≤ 10
  * Major burn (˃30% body surface area)
  * Major trauma requiring ICU admission
  * Spinal cord injury requiring ICU admission

If patient has two or more of the following:

* Administration of ˃ 100 mg daily of prednisolone (or equivalent)
* Sepsis
* Acute renal failure
* Acute hepatic failure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥18 years ICU location status stress ulcer prophylaxis in ICU patients when it is no longer indicated according to pre-defined criteria.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-05-13 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
compare the incidence of overt GI bleeds | 24 hours
  To compare the incidence of overt GI bleeds (defined as hematemesis, bloody nasogastric tube aspirate, or melena) between patients who were on stress ulcer prophylaxis versus patients whose acid suppression therapy was discontinued through the stress ulcer prophylaxis minimization protocol.

SECONDARY OUTCOMES:
Identify the acid suppressive therapy reorder rate | 24 hours
  To Identify the acid suppressive therapy reorder frequency
Number of doses avoided | 24 hours
  Number of acid suppressive therapy doses avoided
Incidences of hospital acquired pneumonia (HAP) | 24 hours
  Number of HAP cases occurring
Incidences of C.Difficile infection | 24 hours
  Number of cases of C.Difficile infections occurring
ICU length of stay | 24 hours
  The time frame of ICU stay
incidence of ICU delirium | 24 hours
  number of cases with ICU Delirium
type of pharmacologic agent used | 24 hours
  Different types of medications used
number of patients with clinically important GI bleeding | 24 hours
  Bleeding defined as overt GI bleeding plus one or more of the following within 24 hours such as decrease in systolic pressure, mean arterial pressure or diastolic pressure, orthostatic hypotension or postural tachycardia , drop in hemoglobin, received transfusions of packed red blood cells or need for vasopressors or invasive interventions like endoscopy.
number of discharge prescriptions for acid suppressive therapy | 24 hours
  number of patients getting discharged with acid suppressive therapy

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Michaels, PharmD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Richardson Medical Center, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data or any protected health information will not be shared with anyone that is not delegated to the study. The PI is committed to disseminate research results in a timely fashion. Sharing of results generated by the data analysis during the course of the project will be through presentation at national scientific meetings and/or publication in open access journals. All information obtained will be source de-identified and presented on a large scale and not traceable to any one particular individual.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 3 years
Access Criteria: Clinical Research Institute

REFERENCES:
- [Background] Cook D, Guyatt G. Prophylaxis against Upper Gastrointestinal Bleeding in Hospitalized Patients. N Engl J Med. 2018 Jun 28;378(26):2506-2516. doi: 10.1056/NEJMra1605507. No abstract available. PMID 29949497
- [Background] Cook DJ, Fuller HD, Guyatt GH, Marshall JC, Leasa D, Hall R, Winton TL, Rutledge F, Todd TJ, Roy P, et al. Risk factors for gastrointestinal bleeding in critically ill patients. Canadian Critical Care Trials Group. N Engl J Med. 1994 Feb 10;330(6):377-81. doi: 10.1056/NEJM199402103300601. PMID 8284001
- [Background] ASHP Therapeutic Guidelines on Stress Ulcer Prophylaxis. ASHP Commission on Therapeutics and approved by the ASHP Board of Directors on November 14, 1998. Am J Health Syst Pharm. 1999 Feb 15;56(4):347-79. doi: 10.1093/ajhp/56.4.347. No abstract available. PMID 10690219
- [Background] 4. Guillamondegui OD, et al. Practice management guidelines for stress ulcer prophylaxis. Eastern Association for the Surgery of Trauma (EAST); 2008.
- [Background] Saeed M, Bass S, Chaisson NF. Which ICU patients need stress ulcer prophylaxis? Cleve Clin J Med. 2022 Jul 1;89(7):363-367. doi: 10.3949/ccjm.89a.21085. PMID 35777844
- [Background] Kantorova I, Svoboda P, Scheer P, Doubek J, Rehorkova D, Bosakova H, Ochmann J. Stress ulcer prophylaxis in critically ill patients: a randomized controlled trial. Hepatogastroenterology. 2004 May-Jun;51(57):757-61. PMID 15143910
- [Background] Marik PE, Vasu T, Hirani A, Pachinburavan M. Stress ulcer prophylaxis in the new millennium: a systematic review and meta-analysis. Crit Care Med. 2010 Nov;38(11):2222-8. doi: 10.1097/CCM.0b013e3181f17adf. PMID 20711074
- [Background] Selvanderan SP, Summers MJ, Finnis ME, Plummer MP, Ali Abdelhamid Y, Anderson MB, Chapman MJ, Rayner CK, Deane AM. Pantoprazole or Placebo for Stress Ulcer Prophylaxis (POP-UP): Randomized Double-Blind Exploratory Study. Crit Care Med. 2016 Oct;44(10):1842-50. doi: 10.1097/CCM.0000000000001819. PMID 27635481
- [Background] Ogasawara O, Kojima T, Miyazu M, Sobue K. Impact of the stress ulcer prophylactic protocol on reducing the unnecessary administration of stress ulcer medications and gastrointestinal bleeding: a single-center, retrospective pre-post study. J Intensive Care. 2020 Jan 16;8:10. doi: 10.1186/s40560-020-0427-8. eCollection 2020. PMID 31988751
- [Background] 11. Dhand, ND, Khatkar MS (2014). Statulator: An online statistical calculator. Sample Size Calculator for Comparing Two Independent Proportions. Accessed 16 March 2023 at http://statulator.com/SampleSize/ss2P.html.